CLINICAL TRIAL: NCT04136938
Title: Impact of Social Marketing in Collective Prevention Actions : Case of Fall Prevention Workshop Among Elderly Living in Three French Departments.
Brief Title: Social Marketing in Prevention Actions
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Crédit Agricole Loire / Haute-Loire (Unknown); Jean Monnet University (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN622019/CHUSTE
Record Dates: First submitted 2019-10-18; First posted 2019-10-23 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Sedentary Behavior; Aging
Keywords: Fall; Seniors; Physical activity; Prevention
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group (social marketing campaign): People aged 60 and over will be included. They will receive a social marketing campaign.
  Interventions: Other: Social marketing campaign
- Control group: People aged 60 and over will be included.

INTERVENTIONS:
Other: Social marketing campaign — A social marketing campaign of prevention workshop sessions will be performed.
  Groups: Intervention group (social marketing campaign)

SUMMARY:
Physical Activity (PA) is recognized as the most effective method to prevent falls in the elderly. Yet despite there being a consensus now that Physical Activity (PA) is effective in practice, there remain many obstacles to participation and attendance resulting in Physical Activity (PA) approaches designed to prevent falls actually only benefiting a limited number of elderly subjects. Social marketing has already shown its utility in the construction of prevention programs.

DETAILED DESCRIPTION:
This study uses the social marketing approach to improve a fall prevention program. The intervention territory will receive social marketing campaign while the territory controls will not have a campaign.

The main goal is to improve attendance at our fall prevention program.

ELIGIBILITY:
Inclusion Criteria:

* People living in the one of the territories of the study
* People without medical contraindications to participate in moderate physical activity
* People who has received information about the study and its rights to its data

Exclusion Criteria:

* People unable to attend workshops
* People already registered for adapted physical activity
* People who refused to participate to the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People aged 60 and over.
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of attendance rate of participants at social marketing campaign (%) | Years: 1
  Comparison rate of attendance rate of participants at prevention workshop sessions (%) between interventional and control group.

SECONDARY OUTCOMES:
Rate of attendance rate of participants at fall prevention workshop sessions (%) | Years: 1
  Comparison rate of attendance rate of participants at prevention workshop sessions (%) between interventional and control group.
Life quality of participants measured by SF-36 questionnaire score | Years: 0, 1
  The SF-36 is a self-questionnaire to assess the quality of life and contains 36 items with minimum score 0 (bad quality life) and maximum score at 100 (good quality life).
Physical activity level of participants measured by IPAQ questionnaire | Years: 0, 1
  The International Physical Activity Questionnaire (IPAQ): short version for elderly people is a self-questionnaire to assess the Physical Activity and contains 7 items. Computation of the total score for the short form requires summation of the duration (in minutes) and frequency (days) of walking, moderate-intensity and vigorous-intensity activities.

CONTACTS AND LOCATIONS:
Overall Officials: Luc GOETHALS, PhD student, Principal Investigator — Jean Monnet University
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goethals L, Barth N, Hupin D, Chapoton B, Guyot J, Celarier T, Roche F, Gallopel-Morvan K, Bongue B. Social Marketing Intervention to Engage Older Adults in Balance Workshops for Fall Prevention: A Multicenter Quasi-Experimental Protocol Study. Front Public Health. 2021 Jul 14;9:614119. doi: 10.3389/fpubh.2021.614119. eCollection 2021. PMID 34336750